CLINICAL TRIAL: NCT01227590
Title: Pharmacokinetic Interactions Between an Herbal Medicine (African Potato) and Antiretroviral Agents (Lopinavir/Ritonavir)
Acronym: AP6142
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2629-34853
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Drug Interactions; Human Immunodeficiency Virus
Keywords: Herbal medicine; African Potato; Hypoxis obtusa; Drug interaction; HIV Infections; Acquired Immunodeficiency Syndrome; Healthy Subjects; Anti-retroviral Agents; Lopinavir; Ritonavir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — lopinavir-ritonavir drug combination; Lopinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmacokinetics single-arm (Experimental): The baseline PK of LPV/r will be established after 14 days of taking LPV/r at a dose of 400/100 mg twice daily. This will be followed by a 7 day course of LPV/r and AP together. The AP dose to be administered will be 15 mg/kg/day of hypoxoside.
  Interventions: Drug: Kaletra (lopinavir/ritonavir), African Potato (hypoxis obtusa)

INTERVENTIONS:
Drug: Kaletra (lopinavir/ritonavir), African Potato (hypoxis obtusa) — The baseline PK of LPV/r will be established after 14 days of taking LPV/r at a dose of 400/100 mg twice daily. This will be followed by a 7 day course of LPV/r and AP together. The AP dose to be administered will be 15 mg/kg/day of hypoxoside.

SUMMARY:
The study is being conducted to evaluate whether African potato, an herbal medicine, can be used together with anti-HIV medicines without affecting the amounts of the anti-HIV medicines in the blood. African potato is an African herbal medicine widely used in Africa, particularly sub-Saharan Africa. Although it has not been proven, it is believed to help boost the immune system. Similar studies have been done on herbal medicines especially those that are used in developing countries. In some cases, the herbal treatments can affect the blood levels of other medicines when the medicines are used together. This study will measure the effect of African potato on lopinavir/ritonavir (Kaletra®), a common anti-HIV medicine. Lopinavir/ritonavir is approved by the United States Food and Drug Administration (FDA). The information obtained from this study will tell us if African potato and anti-HIV treatments can be used together to treat HIV infected patients in Africa and other resource poor regions.

ELIGIBILITY:
Inclusion Criteria:

* Absence of HIV infection prior to study entry.
* Male or female aged 18-60 who are able to provide informed consent.
* Subject is within 20%(+/-) of ideal body weight and must weigh at least 550kg
* Healthy subjects without evidence of acute or chronic illness including diabetes, hypertension, CAD, psychiatric illnesses, renal or hepatic impairment.
* Screening laboratory tests that are normal or deemed not clinically significant by the study physician
* Female subjects of childbearing potential must not be pregnant or lactating, must have a negative pregnancy test at screening and must be practicing an adequate method of birth control. Acceptable methods of birth control include use of an intrauterine device (IUD), oral, implanted or injected contraceptives, and barrier methods with spermicide.
* Subjects must sign an informed consent that complies with US Regulations (US 21 CFR 50) and the International Conference on Harmonization (ICH) guidelines prior to undergoing any study-related procedures.
* Subjects agreed to abstain from consuming grapefruit or its juice for at least 48 hours prior to dosing and throughout the study period until the last blood samples were being obtained.
* Subjects agreed to abstain from consuming alcohol /alcoholic beverages for at least 24 hours prior to dosing and throughout the study period until the last blood sample were being obtained.
* Subjects agreed to abstain from use of cigarettes and tobacco products for at least 24 hours prior to dosing and throughout the study period until the last blood samples were being obtained.
* Subjects who agreed to be available for the entire study period and had the ability to understand and communicate with the investigators and staff.

Exclusion Criteria:

* Use of illicit drugs or alcohol that could interfere with the completion of the study.
* Use of any over- the- counter or prescribed drugs unless approved by the principal investigator or study physician.
* Use of drugs that are known to inhibit/ induce CYP450 isozymes or are substrates of CYP3A4, CYP2D6, CYP2C8 enzymes. (use of hormonal contraceptives is permitted except for oral contraceptives)
* Pregnant or breast- feeding.
* History of acute or chronic illnesses, such as diabetes, hypertension, CAD, psychiatric illnesses, renal or hepatic impairment.
* Evidence of acute illness.
* Family history of congenital prolongation of QTc interval or with any conditions known to prolong QTc interval, such as cardiac arrhythmias, bradycardia or severe heart disease
* History of hypokalemia, hypomagnesemia or hypercholesteremia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic drug interaction study to evaluate the effects of African potato(hypoxis obtusa) on the PK of lopinavir/ritonavir. | 35 days
  The study is to evaluate the effects of African Potato (hypoxis obtusa) on the steady state PK of lopinavir/ritonavir by measurement of the PK parameters of LPV/r in presence and absence of AP in healthy volunteers. The baseline PK of LPV/r will be established after 14 days of taking LPV/r at a dose of 400/100 mg twice daily. This will be followed by a 7 day course of LPV/r and hypoxoside (15 mg/kg/day) together. PK analysis of LPV/r will be repeated following the 7 days of co-administration. Each subject will act as their own control.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca T Aweeka, Pharm.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States